CLINICAL TRIAL: NCT07158190
Title: Evaluation of T-cell Responses After Vaccination With the Attenuated Tetravalent Dengue Vaccine (Takeda).
Acronym: RIMVADE
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6832
Record Dates: First submitted 2024-06-25; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Dengue
Keywords: Vaccination; T cell response
MeSH Terms: conditions — Dengue | interventions — Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — n.1 sample of 10-15 mL of whole blood (lithium-heparin and/or EDTA tubes) for the isolation of mononuclear cells (PBMC). n.1 sample in serum tube (4-6 ml).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 30 volunteers: Individuals who have never contracted the dengue infection and individuals who have previously been confirmed dengue seropositive through laboratory analysis.
  Interventions: Biological: Vaccine

INTERVENTIONS:
Biological: Vaccine — Vaccine TAK003 administration

SUMMARY:
Dengue is one of the most epidemiologically and clinically relevant arboviral diseases, affecting half of the global population. This disease is caused by one of the four serotypes of the dengue virus (DENV1-4), belonging to the flavivirus family transmitted to humans by Aedes aegypti and Aedes albopictus mosquitoes. Dengue is not endemic in Europe, and recorded cases are almost exclusively imported by individuals who have recently visited endemic areas. In Italy, several imported cases are recorded every year, although in the past summer season of 2023, numerous autochthonous cases of dengue were observed, with a particular incidence in Rome and Lazio. In 75-80% of cases the first infection is asymptomatic or paucisymptomatic, while in 20-25% of cases flu-like symptoms may appear, in more severe cases, dengue hemorrhagic fever may occur. Individuals who are infected for the first time are protected for life from that particular serotype that caused the infection. However, Individuals who are infected for the second time with a different serotype are at greater risk of severe dengue.To reduce the risk of dengue epidemics, the most effective method is a systematic and continuous mosquito control. Although the use of an effective vaccine remains a primary prevention measure that should be integrated into the healthcare system. The recent vaccine developed, TAK-003, is an innovative live attenuated vaccine based on serotype 2 (DENV-2), which uses recombinant technology to ensure immunization against all four virus serotypes. However, it showed the highest efficacy against DENV-2, both in seropositive and seronegative people.

To date, there is partial knowledge of the dynamics between viral and host factors that influence the development of disease caused by DENV. In this infections it has been observed that T lymphocytes play a crucial role in dealing with viral pathogens with both harmful and beneficial effects. A debate still persists as whether memory T lymphocytes play solely a protective role in secondary DENV infections or may instead have the potential to contribute to immunopathological mechanisms leading to severe forms of dengue.

Our study aims are to investigate the responses of T lymphocytes against DENV, identifying reliable and meaningful markers of protection. This will be achieved by analyzing the response of T lymphocytes to DENV1-4 serotype epitopes in subjects who will be vaccinated with the attenuated tetravalent dengue TAK003.

DETAILED DESCRIPTION:
Inclusion criteria:

Women/Men aged between 18 and 65 years old; generally in good health, confirmed through a medical history questionnaire and basic laboratory tests; availability for the duration of the study, approximately 26 weeks after vaccination; willingness to sign an informed consent form, acknowledging understanding of the objectives, procedures, and risks associated with the study.

Exclusion criteria:

current pregnancy or breastfeeding; recent hospitalization or serious illness in the past four weeks; evidence of clinically significant neurological, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease based on medical history, physical examination, and/or laboratory studies; behavioral, cognitive, or psychiatric disorders that, in the opinion of the investigator, impact the participant's ability to understand and comply with the study protocol; laboratory values of grade 1 or higher for absolute neutrophil count (ANC), alanine aminotransferase (ALT), and serum creatinine as defined in the protocol; any other condition that, in the opinion of the investigator, could compromise participant safety or rights in the study or make the participant unable to follow the protocol; significant alcohol or drug abuse in the past 12 months resulting in medical, occupational, or family problems, as indicated by the participant's history; history of severe allergic reaction or anaphylaxis; severe asthma (emergency room visit or hospitalization in the past 6 months); current viral infection; use of anticoagulant medications; use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 42 days before or after vaccination. Immunosuppressive dose of corticosteroids is defined as equal to or greater than 10 mg of prednisone equivalent per day for equal to or greater than 14 days; receipt of a live vaccine within 28 days or an inactivated vaccine within 14 days prior to vaccination, or expected receipt of any vaccine within 42 days after vaccination; asplenia; receipt of blood products in the past 6 months, including transfusions or immunoglobulins, or expected receipt of any blood product or immunoglobulin within 42 days after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Women/Men aged between 18 and 65 years old; generally in good health, confirmed through a medical history questionnaire and basic laboratory tests;
* availability for the duration of the study, approximately 26 weeks after vaccination;
* willingness to sign an informed consent form, acknowledging understanding of the objectives, procedures, and risks associated with the stud

Exclusion Criteria:

* current pregnancy or breastfeeding;
* recent hospitalization or serious illness in the past four weeks;
* evidence of clinically significant neurological, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease based on medical history, physical examination, and/or laboratory studies;
* behavioral, cognitive, or psychiatric disorders that, in the opinion of the investigator, impact the participant's ability to understand and comply with the study protocol;
* laboratory values of grade 1 or higher for absolute neutrophil count (ANC), alanine aminotransferase (ALT), and serum creatinine as defined in the protocol;
* any other condition that, in the opinion of the investigator, could compromise participant safety or rights in the study or make the participant unable to follow the protocol;
* significant alcohol or drug abuse in the past 12 months resulting in medical, occupational, or family problems, as indicated by the participant's history;
* history of severe allergic reaction or anaphylaxis;
* severe asthma (emergency room visit or hospitalization in the past 6 months);
* current viral infection;
* use of anticoagulant medications;
* use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 42 days before or after vaccination. Immunosuppressive dose of corticosteroids is defined as equal to or greater than 10 mg of prednisone equivalent per day for equal to or greater than 14 days;
* receipt of a live vaccine within 28 days or an inactivated vaccine within 14 days prior to vaccination, or expected receipt of any vaccine within 42 days after vaccination; asplenia;
* receipt of blood products in the past 6 months, including transfusions or immunoglobulins, or expected receipt of any blood product or immunoglobulin within 42 days after vaccination.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who have never contracted the dengue infection and individuals who have previously been confirmed dengue seropositive through laboratory analysis.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
analysis of antibody titres and T cell | 12 months
  Humoral and cellular immunity to the tetravalent Dengue vaccine (Takeda), assessed through analysis of antibody titers and analysis of T cell responses to epitopes of viral antigens C, E, NS2, NS3, NS4, NS5, prM.

SECONDARY OUTCOMES:
T cell against DENV1-4 | 12months
  correlation between T cell response and antibody tirtrest against DENV1-4
comparison antibody and cell response | 12 months
  comparison between cell and antibody response, among sieropositive and sieronegative subjects.
phenotypical charaterization | 12 months
  phenotypical charaterization of Dengue specific T cell induced by vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Torti, Prof, Principal Investigator — Fondazione Policlinico Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universtiario Agostino Gemelli IRCCS, Rome, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bhatt S, Gething PW, Brady OJ, Messina JP, Farlow AW, Moyes CL, Drake JM, Brownstein JS, Hoen AG, Sankoh O, Myers MF, George DB, Jaenisch T, Wint GR, Simmons CP, Scott TW, Farrar JJ, Hay SI. The global distribution and burden of dengue. Nature. 2013 Apr 25;496(7446):504-7. doi: 10.1038/nature12060. Epub 2013 Apr 7. PMID 23563266
- [Result] Tricou V, Yu D, Reynales H, Biswal S, Saez-Llorens X, Sirivichayakul C, Lopez P, Borja-Tabora C, Bravo L, Kosalaraksa P, Vargas LM, Alera MT, Rivera L, Watanaveeradej V, Dietze R, Fernando L, Wickramasinghe VP, Moreira ED Jr, Fernando AD, Gunasekera D, Luz K, Oliveira AL, Tuboi S, Escudero I, Hutagalung Y, Lloyd E, Rauscher M, Zent O, Folschweiller N, LeFevre I, Espinoza F, Wallace D. Long-term efficacy and safety of a tetravalent dengue vaccine (TAK-003): 4.5-year results from a phase 3, randomised, double-blind, placebo-controlled trial. Lancet Glob Health. 2024 Feb;12(2):e257-e270. doi: 10.1016/S2214-109X(23)00522-3. PMID 38245116
- [Result] Tian Y, Sette A, Weiskopf D. Cytotoxic CD4 T Cells: Differentiation, Function, and Application to Dengue Virus Infection. Front Immunol. 2016 Dec 7;7:531. doi: 10.3389/fimmu.2016.00531. eCollection 2016. PMID 28003809